CLINICAL TRIAL: NCT01172821
Title: A Phase III Randomised, Double-blind, Placebo-controlled, Parallel-group Trial to Evaluate Efficacy and Safety of Tiotropium Inhalation Solution Delivered Via Respimat® Inhaler (2.5 and 5 µg Once Daily) Compared With Placebo and Salmeterol HFA MDI (50 µg Twice Daily) Over 24 Weeks in Moderate Persistent Asthma
Brief Title: Evaluation of Tiotropium 2.5 and 5 mcg Once Daily Delivered Via the Respimat® Inhaler Compared to Placebo and Salmeterol HydroFluoroAlkane (HFA) Metered Dose Inhaler (MDI) (50 mcg Twice Daily) in Patient With Moderate Persistent Asthma II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205.419; 2009-018005-43 (EudraCT Number: EudraCT)
Record Dates: First submitted 2010-07-26; First posted 2010-07-30 (Estimated); Results first posted 2014-02-07 (Estimated); Last update posted 2014-06-09 (Estimated); Status verified 2014-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

ARMS (4):
- tiotropium low dose (Experimental): Once daily, delivered with Respimat® inhaler (+ inhalation of placebo HFA MDI twice daily)
  Interventions: Drug: placebo; Drug: tiotropium Respimat® low dose
- tiotropium high dose (Experimental): Once daily, delivered with Respimat® inhaler (+ inhalation of placebo HFA MDI twice daily)
  Interventions: Drug: tiotropium Respimat® high dose; Drug: placebo
- 50 mcg salmeterol (Active Comparator): Twice daily, delivered with HFA MDI (+ inhalation of placebo Respimat® inhaler once daily)
  Interventions: Drug: placebo; Drug: 50 mcg salmeterol HFA MDI
- placebo (Placebo Comparator): Once daily, delivered with Respimat® inhaler + twice daily delivered with HFA MDI
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: placebo — Placebo that represents BI drug
  Arms: placebo
Drug: placebo — Placebo that represents comparator
  Arms: tiotropium low dose
Drug: placebo — Placebo that represents comparator
  Arms: placebo
Drug: tiotropium Respimat® low dose — IMP
  Arms: tiotropium low dose
Drug: placebo — Placebo that represents BI drug
  Arms: 50 mcg salmeterol
Drug: tiotropium Respimat® high dose — IMP
  Arms: tiotropium high dose
Drug: 50 mcg salmeterol HFA MDI — Active comparator
  Arms: 50 mcg salmeterol
Drug: placebo — Placebo that represents comparator
  Arms: tiotropium high dose

SUMMARY:
The aim of this trial is to evaluate the efficacy and safety of 2.5 and 5 mcg tiotropium over a 24-week treatment period as compared to placebo and salmeterol (50 mcg twice daily). Tiotropium inhalation solution delivered by the Respimat® inhaler will be examined on top of maintenance treatment with inhaled corticosteroid controller medication in patients with moderate persistent asthma. Efficacy and safety will be assessed by measuring effects on lung function, effects on asthma exacerbations, effects on quality of life, effects on asthma control, effects on health care resource utilisation, and number of adverse events.

ELIGIBILITY:
Inclusion criteria:

1. All patients must sign and date an Informed Consent Form consistent with International Conference on Harmonisation - Good Clinical Practice (ICH-GCP) guidelines and local legislation prior to participation in the trial (i.e. prior to any trial procedures, including any pre-trial washout of medications and medication restrictions for pulmonary function test at Visit 1).
2. Male or female patients aged at least 18 years but not more than 75 years.
3. All patients must have at least a 3 month history of asthma at the time of enrolment into the trial. The diagnosis should be confirmed at Visit 1 by fulfilling inclusion criterion 5.
4. The initial diagnosis of asthma must have been made before the patient's age of 40.
5. The diagnosis of asthma has to be confirmed at Visit 1 with a bronchodilator reversibility (15 minutes after 400 mcg salbutamol (albuterol)) resulting in a Forced Expiratory Volume in one second (FEV1) increase of at least 12% and at least 200mL.
6. All patients must have been on maintenance treatment with a medium, stable dose of inhaled corticosteroids for at least for 4 weeks prior to Visit 1. 7. All patients must be symptomatic at Visit 1 (screening) and prior to randomisation at Visit 2 as defined by an Asthma Control Questionnaire (ACQ) mean score of at least 1.5.

8. All patients must have a pre-bronchodilator FEV1 at least 60% and less than or equal to 90% of predicted normal at Visit 1.

9. Variation of absolute FEV1 values of Visit 1 (pre-bronchodilator) as compared to Visit 2 (pre-dose) must be within ± 30%.

10. Patients must be never-smokers or ex-smokers who stopped smoking at least one year prior to enrolment (Visit 0) and who have a smoking history of less than 10 pack years.

11. Patients must be able to use the Respimat® inhaler and metered dose inhaler correctly.

12. Patients must be able to perform all trial related procedures including technically acceptable pulmonary function tests and use of electronic diary/peak flow meter.

Exclusion criteria:

1. Patients with a significant disease other than asthma. A significant disease is defined as a disease which, in the opinion of the investigator, may (i) put the patient at risk because of participation in the trial, or (ii) influence the results of the trial, or (iii) cause concern regarding the patient's ability to participate in the trial.
2. Patients with a clinically relevant abnormal screening (Visit 1) haematology or blood chemistry if the abnormality defines a significant disease as defined in exclusion criterion 1.
3. Patients with a recent history (i.e. six months or less) of myocardial infarction.
4. Patients who have been hospitalised for cardiac failure during the past year.
5. Patients with any unstable or life-threatening cardiac arrhythmia or cardiac arrhythmia requiring intervention or a change in drug therapy within the past year.
6. Patients with lung diseases other than asthma (e.g. Chronic Obstructive Pulmonary Disease (COPD)).
7. Patients with known active tuberculosis.
8. Patients with malignancy for which the patient has undergone resection, radiation therapy or chemotherapy within the last five years. Patients with treated basal cell carcinoma are allowed.
9. Patients who have undergone thoracotomy with pulmonary resection. Patients with a history of thoracotomy for other reasons should be evaluated as per exclusion criterion no. 1.
10. Patients with significant alcohol or drug abuse within the past two years.
11. Patients who are currently in a pulmonary rehabilitation program or have completed a pulmonary rehabilitation program in the 6 weeks prior to Visit 1 (screening).
12. Patients with known hypersensitivity to anticholinergic drugs, benzalkonium chloride (BAC), ethylenediamineteraacetic acid (EDTA), salmeterol xinafoate or any other components of the study medication delivery systems.
13. Pregnant or nursing woman.
14. Women of childbearing potential not using a highly effective method of birth control.
15. Patients who have taken an investigational drug within four weeks prior to Visit 1.
16. Patients who have been treated with beta-blocker medication within four weeks prior to Visit 1 and/or during the screening period. Topical cardio-selective beta-blocker eye medications for non-narrow angle glaucoma are allowed.
17. Patients who have been treated with the long-acting anticholinergic tiotropium (Spiriva®) within four weeks prior to Visit 1 and/or during the screening period.
18. Patients who have been treated with oral or patch beta-adrenergics within four weeks prior to Visit 1 and/or during the Screening period.
19. Patients who have been treated with oral corticosteroids within four weeks prior to Visit 1 and/or during the screening period.
20. Patients who have been treated with anti-IgE antibodies, e.g. omalizumab (Xolair®), within 6 months prior to Visit 1 and/or during the screening period.
21. Patients who have been treated with cromone within two weeks prior to Visit 1 and/or during the screening period.
22. Patients who have been treated with methylxanthines or phosphodiesterase 4 inhibitors within two weeks prior to Visit 1 and/or during the screening period.
23. Patients who have been treated with other non-approved and according to international guidelines not recommended "experimental" drugs for routine asthma therapy within four weeks prior to Visit 1 and/or during the screening period.
24. Patients with any asthma exacerbation or any respiratory tract infection iin the four weeks prior to Visit 1 and/or during the screening period.
25. Patients who have previously been randomised in this trial or in the respective twin trial (205.418) or are currently participating in another trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1032 (Actual)
Dates: Start 2010-08; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (125):
- United States (18):
  - 205.419.01058 Boehringer Ingelheim Investigational Site, Los Angeles, California
  - 205.419.01053 Boehringer Ingelheim Investigational Site, Stockton, California
  - 205.419.01061 Boehringer Ingelheim Investigational Site, Centennial, Colorado
  - 205.419.01066 Boehringer Ingelheim Investigational Site, Denver, Colorado
  - 205.419.01064 Boehringer Ingelheim Investigational Site, Panama City, Florida
  - 205.419.01060 Boehringer Ingelheim Investigational Site, Winter Park, Florida
  - 205.419.01068 Boehringer Ingelheim Investigational Site, Novi, Michigan
  - 205.419.01054 Boehringer Ingelheim Investigational Site, Plymouth, Minnesota
  - 205.419.01062 Boehringer Ingelheim Investigational Site, St Louis, Missouri
  - 205.419.01070 Boehringer Ingelheim Investigational Site, Bozeman, Montana
  - 205.419.01067 Boehringer Ingelheim Investigational Site, Skillman, New Jersey
  - 205.419.01071 Boehringer Ingelheim Investigational Site, Raleigh, North Carolina
  - 205.419.01055 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 205.419.01065 Boehringer Ingelheim Investigational Site, Portland, Oregon
  - 205.419.01069 Boehringer Ingelheim Investigational Site, Greenville, South Carolina
  - 205.419.01056 Boehringer Ingelheim Investigational Site, Union, South Carolina
  - 205.419.01063 Boehringer Ingelheim Investigational Site, El Paso, Texas
  - 205.419.01051 Boehringer Ingelheim Investigational Site, San Antonio, Texas
- Brazil (4):
  - 205.419.55053 Boehringer Ingelheim Investigational Site, Florianópolis
  - 205.419.55054 Boehringer Ingelheim Investigational Site, Porto Alegre
  - 205.419.55052 Boehringer Ingelheim Investigational Site, São Paulo
  - 205.419.55055 Boehringer Ingelheim Investigational Site, São Paulo
- China (17):
  - 205.419.86061 Boehringer Ingelheim Investigational Site, Chengdu
  - 205.419.86053 Boehringer Ingelheim Investigational Site, Chongqing
  - 205.419.86056 Boehringer Ingelheim Investigational Site, Guangzhou
  - 205.419.86062 Boehringer Ingelheim Investigational Site, Guangzhou
  - 205.419.86054 Boehringer Ingelheim Investigational Site, Haikou
  - 205.419.86059 Boehringer Ingelheim Investigational Site, Kunming
  - 205.419.86058 Boehringer Ingelheim Investigational Site, Nanchang
  - 205.419.86064 Boehringer Ingelheim Investigational Site, Nanjing
  - 205.419.86051 Boehringer Ingelheim Investigational Site, Shanghai
  - 205.419.86052 Boehringer Ingelheim Investigational Site, Shanghai
  - 205.419.86055 Boehringer Ingelheim Investigational Site, Shanghai
  - 205.419.86066 Boehringer Ingelheim Investigational Site, Shanghai
  - 205.419.86057 Boehringer Ingelheim Investigational Site, Xi'an
  - 205.419.86065 Boehringer Ingelheim Investigational Site, Xi'an
  - 205.419.86063 Boehringer Ingelheim Investigational Site, Xuzhou
  - 205.419.86067 Boehringer Ingelheim Investigational Site, Yangzhou
  - 205.419.86068 Boehringer Ingelheim Investigational Site, Yinchuan
- Colombia (4):
  - 205.419.57051 Boehringer Ingelheim Investigational Site, Bogotá
  - 205.419.57052 Boehringer Ingelheim Investigational Site, Bogotá
  - 205.419.57053 Boehringer Ingelheim Investigational Site, Bogotá
  - 205.419.57054 Boehringer Ingelheim Investigational Site, Medellín
- Germany (13):
  - 205.419.49061 Boehringer Ingelheim Investigational Site, Bamberg
  - 205.419.49051 Boehringer Ingelheim Investigational Site, Berlin
  - 205.419.49052 Boehringer Ingelheim Investigational Site, Berlin
  - 205.419.49062 Boehringer Ingelheim Investigational Site, Berlin
  - 205.419.49063 Boehringer Ingelheim Investigational Site, Berlin
  - 205.419.49064 Boehringer Ingelheim Investigational Site, Berlin
  - 205.419.49054 Boehringer Ingelheim Investigational Site, Frankfurt
  - 205.419.49058 Boehringer Ingelheim Investigational Site, Hamburg
  - 205.419.49057 Boehringer Ingelheim Investigational Site, Koblenz
  - 205.419.49056 Boehringer Ingelheim Investigational Site, Lübeck
  - 205.419.49059 Boehringer Ingelheim Investigational Site, Rüdersdorf
  - 205.419.49053 Boehringer Ingelheim Investigational Site, Wiesbaden
  - 205.419.49055 Boehringer Ingelheim Investigational Site, Witten
- India (8):
  - 205.419.91057 Boehringer Ingelheim Investigational Site, Ahmedabad
  - 205.419.91056 Boehringer Ingelheim Investigational Site, Coimbatore
  - 205.419.91055 Boehringer Ingelheim Investigational Site, Hyderabad
  - 205.419.91051 Boehringer Ingelheim Investigational Site, Jaipur
  - 205.419.91058 Boehringer Ingelheim Investigational Site, Jaipur
  - 205.419.91054 Boehringer Ingelheim Investigational Site, Mumbai
  - 205.419.91059 Boehringer Ingelheim Investigational Site, Mysore
  - 205.419.91053 Boehringer Ingelheim Investigational Site, Nagpur
- Japan (35):
  - 205.419.81085 Boehringer Ingelheim Investigational Site, Aira, Kagoshima
  - 205.419.81062 Boehringer Ingelheim Investigational Site, Chuo-ku, Tokyo
  - 205.419.81073 Boehringer Ingelheim Investigational Site, Fukuoka, Fukuoka
  - 205.419.81074 Boehringer Ingelheim Investigational Site, Fukuoka, Fukuoka
  - 205.419.81072 Boehringer Ingelheim Investigational Site, Fukuyama, Hiroshima
  - 205.419.81069 Boehringer Ingelheim Investigational Site, Habikino, Osaka
  - 205.419.81071 Boehringer Ingelheim Investigational Site, Hiroshima, Hiroshima
  - 205.419.81058 Boehringer Ingelheim Investigational Site, Itabashi-ku, Tokyo
  - 205.419.81064 Boehringer Ingelheim Investigational Site, Iwata, Shizuoka
  - 205.419.81063 Boehringer Ingelheim Investigational Site, Kanazawa, Ishikawa
  - 205.419.81054 Boehringer Ingelheim Investigational Site, Kishiwada, Osaka
  - 205.419.81075 Boehringer Ingelheim Investigational Site, Kitakyushu, Fukuoka
  - 205.419.81070 Boehringer Ingelheim Investigational Site, Kobe, Hyogo
  - 205.419.81061 Boehringer Ingelheim Investigational Site, Koto-ku, Tokyo
  - 205.419.81067 Boehringer Ingelheim Investigational Site, Kyoto, Kyoto
  - 205.419.81080 Boehringer Ingelheim Investigational Site, Matsusaka, Mie
  - 205.419.81081 Boehringer Ingelheim Investigational Site, Meguro-ku, Tokyo
  - 205.419.81060 Boehringer Ingelheim Investigational Site, Minato-ku, Tokyo
  - 205.419.81077 Boehringer Ingelheim Investigational Site, Minato-ku, Tokyo
  - 205.419.81056 Boehringer Ingelheim Investigational Site, Morioka, Iwate
  - 205.419.81055 Boehringer Ingelheim Investigational Site, Naka-gun, Ibaraki
  - 205.419.81078 Boehringer Ingelheim Investigational Site, Nakano-ku,Tokyo
  - 205.419.81084 Boehringer Ingelheim Investigational Site, Oita,Oita
  - 205.419.81068 Boehringer Ingelheim Investigational Site, Osaka-Sayama, Osaka
  - 205.419.81053 Boehringer Ingelheim Investigational Site, Sapporo, Hokkaido
  - 205.419.81057 Boehringer Ingelheim Investigational Site, Sendai, Miyagi
  - 205.419.81059 Boehringer Ingelheim Investigational Site, Seto, Aichi
  - 205.419.81082 Boehringer Ingelheim Investigational Site, Shinagawa-ku, Tokyo
  - 205.419.81065 Boehringer Ingelheim Investigational Site, Shizuoka, Shizuoka
  - 205.419.81066 Boehringer Ingelheim Investigational Site, Toyota, Aichi
  - 205.419.81051 Boehringer Ingelheim Investigational Site, Urasoe, Okinawa
  - 205.419.81052 Boehringer Ingelheim Investigational Site, Urasoe, Okinawa
  - 205.419.81076 Boehringer Ingelheim Investigational Site, Urasoe, Okinawa
  - 205.419.81083 Boehringer Ingelheim Investigational Site, Yokohama, Kanagawa
  - 205.419.81079 Boehringer Ingelheim Investigational Site, Yotsukaido, Chiba
- Mexico (3):
  - 205.419.52051 Boehringer Ingelheim Investigational Site, Mexico City
  - 205.419.52052 Boehringer Ingelheim Investigational Site, Mexico City
  - 205.419.52053 Boehringer Ingelheim Investigational Site, Monterrey
- Peru (5):
  - 205.419.51051 Boehringer Ingelheim Investigational Site, Lima
  - 205.419.51052 Boehringer Ingelheim Investigational Site, Lima
  - 205.419.51053 Boehringer Ingelheim Investigational Site, Lima
  - 205.419.51054 Boehringer Ingelheim Investigational Site, Lima
  - 205.419.51055 Boehringer Ingelheim Investigational Site, Lima
- Poland (8):
  - 205.419.48052 Boehringer Ingelheim Investigational Site, Bialystok
  - 205.419.48054 Boehringer Ingelheim Investigational Site, Bydgoszcz
  - 205.419.48055 Boehringer Ingelheim Investigational Site, Gorzów Wielkopolski
  - 205.419.48051 Boehringer Ingelheim Investigational Site, Krakow
  - 205.419.48057 Boehringer Ingelheim Investigational Site, Poznan
  - 205.419.48058 Boehringer Ingelheim Investigational Site, Sopot
  - 205.419.48056 Boehringer Ingelheim Investigational Site, Wroclaw
  - 205.419.48053 Boehringer Ingelheim Investigational Site, Włoszczowa
- Romania (10):
  - 205.419.40055 Boehringer Ingelheim Investigational Site, Brasov
  - 205.419.40056 Boehringer Ingelheim Investigational Site, Brasov
  - 205.419.40051 Boehringer Ingelheim Investigational Site, Bucharest
  - 205.419.40052 Boehringer Ingelheim Investigational Site, Bucharest
  - 205.419.40053 Boehringer Ingelheim Investigational Site, Bucharest
  - 205.419.40054 Boehringer Ingelheim Investigational Site, Bucharest
  - 205.419.40058 Boehringer Ingelheim Investigational Site, Bucharest
  - 205.419.40060 Boehringer Ingelheim Investigational Site, Bucharest
  - 205.419.40059 Boehringer Ingelheim Investigational Site, Constanța
  - 205.419.40057 Boehringer Ingelheim Investigational Site, Iași

REFERENCES:
- [Derived] Halpin DMG, Hamelmann EH, Frith PA, Moroni-Zentgraf PM, van Hecke B, Unseld A, Kerstjens HAM, Szefler SJ. Comparative Responses in Lung Function Measurements with Tiotropium in Adolescents and Adults, and Across Asthma Severities: A Post Hoc Analysis. Pulm Ther. 2020 Jun;6(1):131-140. doi: 10.1007/s41030-020-00113-w. Epub 2020 Mar 16. PMID 32180164
- [Derived] Casale TB, Aalbers R, Bleecker ER, Meltzer EO, Zaremba-Pechmann L, de la Hoz A, Kerstjens HAM. Tiotropium Respimat(R) add-on therapy to inhaled corticosteroids in patients with symptomatic asthma improves clinical outcomes regardless of baseline characteristics. Respir Med. 2019 Oct-Nov;158:97-109. doi: 10.1016/j.rmed.2019.09.014. Epub 2019 Sep 30. PMID 31654891
- [Derived] Halpin DMG, Meltzer EO, Pisternick-Ruf W, Moroni-Zentgraf P, Engel M, Zaremba-Pechmann L, Casale T, FitzGerald JM. Peak expiratory flow as an endpoint for clinical trials in asthma: a comparison with FEV1. Respir Res. 2019 Jul 18;20(1):159. doi: 10.1186/s12931-019-1119-6. PMID 31319851
- [Derived] Casale TB, Bateman ED, Vandewalker M, Virchow JC, Schmidt H, Engel M, Moroni-Zentgraf P, Kerstjens HAM. Tiotropium Respimat Add-on Is Efficacious in Symptomatic Asthma, Independent of T2 Phenotype. J Allergy Clin Immunol Pract. 2018 May-Jun;6(3):923-935.e9. doi: 10.1016/j.jaip.2017.08.037. Epub 2017 Nov 22. PMID 29174062
- [Derived] Kerstjens HA, Casale TB, Bleecker ER, Meltzer EO, Pizzichini E, Schmidt O, Engel M, Bour L, Verkleij CB, Moroni-Zentgraf P, Bateman ED. Tiotropium or salmeterol as add-on therapy to inhaled corticosteroids for patients with moderate symptomatic asthma: two replicate, double-blind, placebo-controlled, parallel-group, active-comparator, randomised trials. Lancet Respir Med. 2015 May;3(5):367-76. doi: 10.1016/S2213-2600(15)00031-4. Epub 2015 Feb 12. PMID 25682232

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There was 1 patient in the TIO R2.5 and 1 patient in the TIO R5 group randomized but not treated.
Groups:
- Placebo: Matching Placebo delivered by the Respimat Inhaler resp. MDI (hydrofluoroalkane (HFA 134a) metered inhaler).
- Tio R2.5: Tiotropium 2.5 microgram (mcg) qd (evening) delivered by the Respimat Inhaler.
- Tio R5: Tiotropium 5 mcg qd (evening) delivered by the Respimat Inhaler.
- Salmeterol: Salmeterol 50 mcg bid (morning and evening) delivered by the MDI (hydrofluoroalkane (HFA 134a) metered inhaler).
Period: Overall Study
Arm/Group | Placebo | Tio R2.5 | Tio R5 | Salmeterol
Started | 254 (Entered and Treated) | 257 (Entered and Treated) | 253 (Entered and Treated) | 266 (Entered and Treated)
Completed | 240 | 245 | 240 | 249
Not Completed | 14 | 12 | 13 | 17
Not completed — Adverse Event | 5 | 2 | 2 | 7
Not completed — Protocol Violation | 0 | 2 | 1 | 2
Not completed — Lost to Follow-up | 4 | 1 | 2 | 2
Not completed — Withdrawal by Subject | 2 | 3 | 3 | 3
Not completed — Other | 3 | 4 | 5 | 3

BASELINE CHARACTERISTICS:
Population: Treated Set (TS) - all randomised patients who received at least 1 dose of randomised trial medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Tio R2.5 | Tio R5 | Salmeterol | Total
Number analyzed (Participants) | 254 | 257 | 253 | 266 | 1030
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.0 (13.0) | 43.0 (12.6) | 44.3 (12.7) | 41.5 (13.1) | 42.9 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 145 | 160 | 146 | 153 | 604
  Male | 109 | 97 | 107 | 113 | 426

OUTCOME MEASURES:

1. Primary Outcome: Peak FEV1 Within 3 Hours Post-dose Response
Description: Peak forced expiratory volume in one second (FEV1) response within 3 hours post-dose determined at the end of the 24-week treatment. Response was defined as change from baseline (10 minutes before the first dose of trial medication at visit 2). Means are adjusted for treatment, centre, week, baseline, treatment by week, and baseline by week.
Time Frame: 24 weeks
Population: Full Analysis Set (FAS) - all treated patients who had baseline data and at least 1 on-treatment efficacy measurement.
Measure: Mean (Standard Error); unit: Litre
Arm/Group | Placebo | Tio R2.5 | Tio R5 | Salmeterol
Number analyzed (Participants) | 242 | 245 | 240 | 251
Litre | 0.075 (0.020) | 0.287 (0.020) | 0.244 (0.020) | 0.252 (0.019)
Statistical Analysis 1: Comparison: Placebo vs Tio R2.5; Analyses included the fixed, categorical effects of treatment, centre, week, and treatment-by-week interaction, as well as the covariates of baseline value and baseline value-by-week interaction. Patient was included as a random effect in the model; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Adjusted using a restricted maximum likelihood (REML)-based mixed effects model with repeated measures (MMRM); Mean Difference (Final Values) = 0.211, 95% CI 2-sided [0.159 to 0.264], Standard Error of Mean 0.027 — Tio R2.5 - Placebo
Statistical Analysis 2: Comparison: Placebo vs Tio R5; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Adjusted using a restricted maximum likelihood (REML)-based mixed effects model with repeated measures (MMRM); Mean Difference (Final Values) = 0.169, 95% CI 2-sided [0.116 to 0.222], Standard Error of Mean 0.027 — Tio R5 - Placebo

2. Primary Outcome: Trough FEV1 Response
Description: Trough FEV1 response determined at the end of the 24-week treatment. Response was defined as change from baseline (10 minutes before the first dose of trial medication at visit 2). Means are adjusted for treatment, centre, week, baseline, treatment by week, and baseline by week.
Time Frame: 24 weeks
Population: FAS
Measure: Mean (Standard Error); unit: Litre
Arm/Group | Placebo | Tio R2.5 | Tio R5 | Salmeterol
Number analyzed (Participants) | 242 | 245 | 240 | 251
Litre | -0.012 (0.021) | 0.164 (0.021) | 0.121 (0.021) | 0.094 (0.021)
Statistical Analysis 1: Comparison: Placebo vs Tio R2.5; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Adjusted using a restricted maximum likelihood (REML)-based mixed effects model with repeated measures (MMRM); Mean Difference (Final Values) = 0.176, 95% CI 2-sided [0.120 to 0.233], Standard Error of Mean 0.029 — Tio R2.5 - Placebo
Statistical Analysis 2: Comparison: Placebo vs Tio R5; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Adjusted using a restricted maximum likelihood (REML)-based mixed effects model with repeated measures (MMRM); Mean Difference (Final Values) = 0.133, 95% CI 2-sided [0.076 to 0.190], Standard Error of Mean 0.029 — Tio R5 - Placebo

3. Secondary Outcome: Peak FVC Within 3 Hours Post-dose Response
Description: Peak forced vital capacity (FVC) response within 3 hours post-dose determined at the end of the 24-week treatment. Response was defined as change from baseline (10 minutes before the first dose of trial medication at visit 2). Means are adjusted for treatment, centre, week, baseline, treatment by week, and baseline by week.
Time Frame: 24 weeks
Population: FAS
Measure: Mean (Standard Error); unit: Litre
Arm/Group | Placebo | Tio R2.5 | Tio R5 | Salmeterol
Number analyzed (Participants) | 242 | 245 | 240 | 251
Litre | 0.071 (0.022) | 0.181 (0.022) | 0.160 (0.022) | 0.188 (0.021)
Statistical Analysis 1: Comparison: Placebo vs Tio R2.5; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis; Adjusted using a restricted maximum likelihood (REML)-based mixed effects model with repeated measures (MMRM); Mean Difference (Final Values) = 0.110, 95% CI 2-sided [0.052 to 0.168], Standard Error of Mean 0.030 — Tio R2.5 - Placebo
Statistical Analysis 2: Comparison: Placebo vs Tio R5; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0031, Mixed Models Analysis; Adjusted using a restricted maximum likelihood (REML)-based mixed effects model with repeated measures (MMRM); Mean Difference (Final Values) = 0.089, 95% CI 2-sided [0.030 to 0.147], Standard Error of Mean 0.030 — Tio R5 - Placebo

4. Secondary Outcome: Trough FVC Response
Description: Trough FVC response determined at the end of the 24-week treatment. Response was defined as change from baseline (10 minutes before the first dose of trial medication at visit 2). Means are adjusted for treatment, country, week, baseline, treatment by week, and baseline by week.
Time Frame: 24 weeks
Population: FAS
Measure: Mean (Standard Error); unit: Litre
Arm/Group | Placebo | Tio R2.5 | Tio R5 | Salmeterol
Number analyzed (Participants) | 242 | 245 | 240 | 251
Litre | -0.048 (0.027) | 0.039 (0.027) | 0.035 (0.027) | 0.020 (0.027)
Statistical Analysis 1: Comparison: Placebo vs Tio R2.5; Analyses included the fixed, categorical effects of treatment, country, week, and treatment-by-week interaction, as well as the covariates of baseline value and baseline value-by-week interaction. Patient was included as a random effect in the model; Test type: Superiority or Other; p = 0.0061, Mixed Models Analysis; Adjusted using a restricted maximum likelihood (REML)-based mixed effects model with repeated measures (MMRM); Mean Difference (Final Values) = 0.087, 95% CI 2-sided [0.025 to 0.149], Standard Error of Mean 0.032 — Tio R2.5 - Placebo
Statistical Analysis 2: Comparison: Placebo vs Tio R5; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0093, Mixed Models Analysis; Adjusted using a restricted maximum likelihood (REML)-based mixed effects model with repeated measures (MMRM); Mean Difference (Final Values) = 0.083, 95% CI 2-sided [0.021 to 0.146], Standard Error of Mean 0.032 — Tio R5 - Placebo

5. Secondary Outcome: FEV1 Area Under Curve 0-3 Hours (AUC0-3h) Response
Description: Response was defined as change from baseline (10 minutes before the first dose of trial medication at visit 2) determined at the end of the 24- week treatment. Means are adjusted for treatment, centre, week, baseline, treatment by week, and baseline by week. FEV1 AUC 0-3h was calculated from 0-3 hours post-dose using the trapezoidal rule, divided by the observation time (3h) to report in litres.
Time Frame: 24 weeks
Population: FAS
Measure: Mean (Standard Error); unit: Litre
Arm/Group | Placebo | Tio R2.5 | Tio R5 | Salmeterol
Number analyzed (Participants) | 242 | 245 | 240 | 251
Litre | -0.005 (0.019) | 0.196 (0.019) | 0.158 (0.019) | 0.173 (0.019)
Statistical Analysis 1: Comparison: Placebo vs Tio R2.5; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Adjusted using a restricted maximum likelihood (REML)-based mixed effects model with repeated measures (MMRM); Mean Difference (Final Values) = 0.201, 95% CI 2-sided [0.150 to 0.252], Standard Error of Mean 0.026 — Tio R2.5 - Placebo
Statistical Analysis 2: Comparison: Placebo vs Tio R5; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Adjusted using a restricted maximum likelihood (REML)-based mixed effects model with repeated measures (MMRM); Mean Difference (Final Values) = 0.163, 95% CI 2-sided [0.112 to 0.215], Standard Error of Mean 0.026 — Tio R5 - Placebo

6. Secondary Outcome: FVC Area Under Curve 0-3 Hours (AUC0-3h) Response
Description: Response was defined as change from baseline (10 minutes before the first dose of trial medication at visit 2) determined at the end of the 24- week treatment. Means are adjusted for treatment, country, week, baseline, treatment by week, and baseline by week. FVC AUC 0-3h was calculated from 0-3 hours post-dose using the trapezoidal rule, divided by the observation time (3h) to report in litres.
Time Frame: 24 weeks
Population: FAS
Measure: Mean (Standard Error); unit: Litre
Arm/Group | Placebo | Tio R2.5 | Tio R5 | Salmeterol
Number analyzed (Participants) | 242 | 245 | 240 | 251
Litre | -0.065 (0.024) | 0.043 (0.024) | 0.024 (0.025) | 0.066 (0.024)
Statistical Analysis 1: Comparison: Placebo vs Tio R2.5; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis; Adjusted using a restricted maximum likelihood (REML)-based mixed effects model with repeated measures (MMRM); Mean Difference (Final Values) = 0.108, 95% CI 2-sided [0.052 to 0.164], Standard Error of Mean 0.029 — Tio R2.5 - Placebo
Statistical Analysis 2: Comparison: Placebo vs Tio R5; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0019, Mixed Models Analysis; Adjusted using a restricted maximum likelihood (REML)-based mixed effects model with repeated measures (MMRM); Mean Difference (Final Values) = 0.089, 95% CI 2-sided [0.033 to 0.145], Standard Error of Mean 0.029 — Tio R5 - Placebo

7. Secondary Outcome: Trough PEF Response
Description: Trough peak expiratory flow (PEF) response determined at the end of the 24-week treatment. Response was defined as change from baseline (10 minutes before the first dose of trial medication at visit 2). Means are adjusted for treatment, centre, week, baseline, treatment by week, and baseline by week.
Time Frame: 24 weeks
Population: FAS
Measure: Mean (Standard Error); unit: Litre/min
Arm/Group | Placebo | Tio R2.5 | Tio R5 | Salmeterol
Number analyzed (Participants) | 242 | 245 | 240 | 251
Litre/min | 7.938 (3.659) | 36.698 (3.614) | 36.117 (3.646) | 29.352 (3.572)
Statistical Analysis 1: Comparison: Placebo vs Tio R2.5; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Adjusted using a restricted maximum likelihood (REML)-based mixed effects model with repeated measures (MMRM); Mean Difference (Final Values) = 28.759, 95% CI 2-sided [19.025 to 38.494], Standard Error of Mean 4.963 — Tio R2.5 - Placebo
Statistical Analysis 2: Comparison: Placebo vs Tio R5; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Adjusted using a restricted maximum likelihood (REML)-based mixed effects model with repeated measures (MMRM); Mean Difference (Final Values) = 28.178, 95% CI 2-sided [18.401 to 37.956], Standard Error of Mean 4.985 — Tio R5 - Placebo

8. Secondary Outcome: Total Asthma Quality of Life Questionnaire (AQLQs)) Score
Description: Total score from the Standardised Asthma Quality of Life Questionnaire (AQLQ(s)) determined at the end of 24-week treatment.
  The AQLQ(s) contains 32 questions, each question has a 7 point scale from 1 (highest intensity) till 7 (no symptoms). Total score was defined as the sum of all items divided by the number of items and ranges from from 1 (highest intensity) till 7 (no symptoms). Means are adjusted for treatment, centre, week, baseline, treatment by week, and baseline by week.
Time Frame: 24 weeks
Population: FAS
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tio R2.5 | Tio R5 | Salmeterol
Number analyzed (Participants) | 240 | 245 | 240 | 250
units on a scale | 5.551 (0.050) | 5.562 (0.049) | 5.548 (0.050) | 5.634 (0.048)
Statistical Analysis 1: Comparison: Placebo vs Tio R2.5; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.8700, Mixed Models Analysis; Adjusted using a restricted maximum likelihood (REML)-based mixed effects model with repeated measures (MMRM); Mean Difference (Final Values) = 0.011, 95% CI 2-sided [-0.122 to 0.144], Standard Error of Mean 0.068 — Tio R2.5 - Placebo
Statistical Analysis 2: Comparison: Placebo vs Tio R5; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.9612, Mixed Models Analysis; Adjusted using a restricted maximum likelihood (REML)-based mixed effects model with repeated measures (MMRM); Mean Difference (Final Values) = -0.003, 95% CI 2-sided [-0.137 to 0.130], Standard Error of Mean 0.068 — Tio R5 - Placebo

9. Secondary Outcome: Total Asthma Control Questionnaire (ACQ) Score
Description: Control of asthma as assessed by the ACQ determined at the end of 24-week treatment. The ACQ contains 7 questions, each question has a 7 point scale from 0 (no symptoms) till 6 (highest intensity). Total score was defined as the sum of all items divided by the number of items and ranges from from 0 (no symptoms) till 6 (highest intensity). Means are adjusted for treatment, centre, week, baseline, treatment by week, and baseline by week.
Time Frame: 24 weeks
Population: FAS
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tio R2.5 | Tio R5 | Salmeterol
Number analyzed (Participants) | 240 | 245 | 240 | 250
units on a scale | 1.442 (0.043) | 1.315 (0.042) | 1.359 (0.043) | 1.318 (0.042)
Statistical Analysis 1: Comparison: Placebo vs Tio R2.5; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0305, Mixed Models Analysis; Adjusted using a restricted maximum likelihood (REML)-based mixed effects model with repeated measures (MMRM); Mean Difference (Final Values) = -0.127, 95% CI 2-sided [-0.241 to -0.012], Standard Error of Mean 0.059 — Tio R2.5 - Placebo
Statistical Analysis 2: Comparison: Placebo vs Tio R5; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1602, Mixed Models Analysis; Adjusted using a restricted maximum likelihood (REML)-based mixed effects model with repeated measures (MMRM); Mean Difference (Final Values) = -0.083, 95% CI 2-sided [-0.198 to 0.033], Standard Error of Mean 0.059 — Tio R5 - Placebo

10. Secondary Outcome: The Responder Rate as Assessed by the ACQ
Description: The responder rate as assessed by the Asthma Control Questionnaire (ACQ) determined at the end of the 24-week treatment period. A patient was considered to be a responder if he or she was reported with an improvement (decrease) in ACQ total score of at least 0.5 points.The score ranges from 0 (no impairment) to 6 (maximum impairment).
Time Frame: 24 weeks
Population: FAS
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Tio R2.5 | Tio R5 | Salmeterol
Number analyzed (Participants) | 253 | 256 | 252 | 264
Percentage of participants | 62.5 | 66.4 | 61.9 | 64.4
Statistical Analysis 1: Comparison: Placebo vs Tio R2.5; Test type: Superiority or Other; p = 0.4012, Fisher Exact — Calculated as 2*one-sided-p-value in the direction corresponding to testing the null hypothesis; Odds Ratio (OR) = 1.19, 95% CI 2-sided [0.81 to 1.74] — Tio R2.5 / Placebo
Statistical Analysis 2: Comparison: Placebo vs Tio R5; Test type: Superiority or Other; p = 1.1727, Fisher Exact — Calculated as 2*one-sided-p-value in the direction corresponding to testing the null hypothesis; Odds Ratio (OR) = 0.98, 95% CI 2-sided [0.67 to 1.42] — Tio R5 / Placebo

11. Secondary Outcome: Mean Pre-dose Morning PEF (PEF a.m.) Based on the Weekly Mean Response at Week 24
Description: Weekly means obtained during the last 7 days before week 24 measured by patients at home using the AM3 device. Response was defined as change from baseline. Means are adjusted for treatment, country, week, baseline, treatment by week, and baseline by week
Time Frame: Baseline and last 7 days before week 24 visit
Population: FAS
Measure: Mean (Standard Error); unit: Litre/min
Arm/Group | Placebo | Tio R2.5 | Tio R5 | Salmeterol
Number analyzed (Participants) | 235 | 238 | 236 | 247
Litre/min | 2.764 (3.292) | 23.377 (3.267) | 27.521 (3.294) | 19.779 (3.219)
Statistical Analysis 1: Comparison: Placebo vs Tio R2.5; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Adjusted using a restricted maximum likelihood (REML)-based mixed effects model with repeated measures (MMRM); Mean Difference (Final Values) = 20.613, 95% CI 2-sided [11.795 to 29.431], Standard Error of Mean 4.496 — Tio R2.5 - Placebo
Statistical Analysis 2: Comparison: Placebo vs Tio R5; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Adjusted using a restricted maximum likelihood (REML)-based mixed effects model with repeated measures (MMRM); Mean Difference (Final Values) = 24.757, 95% CI 2-sided [15.907 to 33.607], Standard Error of Mean 4.513 — Tio R5 - Placebo

12. Secondary Outcome: Mean Pre-dose Evening PEF (PEF p.m.) Based on the Weekly Mean Response at Week 24
Description: as for outcome 11
Time Frame: Baseline and last 7 days before week 24 visit
Population: FAS
Measure: Mean (Standard Error); unit: Litre/min
Arm/Group | Placebo | Tio R2.5 | Tio R5 | Salmeterol
Number analyzed (Participants) | 236 | 238 | 236 | 247
Litre/min | -0.072 (3.328) | 15.919 (3.303) | 21.175 (3.330) | 11.617 (3.256)
Statistical Analysis 1: Comparison: Placebo vs Tio R2.5; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0004, Mixed Models Analysis; Adjusted using a restricted maximum likelihood (REML)-based mixed effects model with repeated measures (MMRM); Mean Difference (Final Values) = 15.991, 95% CI 2-sided [7.074 to 24.908], Standard Error of Mean 4.547 — Tio R2.5 - Placebo
Statistical Analysis 2: Comparison: Placebo vs Tio R5; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Adjusted using a restricted maximum likelihood (REML)-based mixed effects model with repeated measures (MMRM); Mean Difference (Final Values) = 21.247, 95% CI 2-sided [12.302 to 30.193], Standard Error of Mean 4.561 — Tio R5 - Placebo

13. Secondary Outcome: PEF Variability
Description: PEF daily variability was assesed by patients at home using the AM3 device. PEF variability is the absolute difference between morning and evening PEF value divided by their mean, based on the weekly mean response at week 24. Means are adjusted for treatment, country, week, baseline, treatment by week, and baseline by week.
Time Frame: Last 7 days before week 24 visit
Population: FAS
Measure: Mean (Standard Error); unit: Percentage of Mean PEF
Arm/Group | Placebo | Tio R2.5 | Tio R5 | Salmeterol
Number analyzed (Participants) | 232 | 237 | 234 | 244
Percentage of Mean PEF | -0.448 (0.484) | -1.401 (0.480) | -0.627 (0.487) | -1.518 (0.472)
Statistical Analysis 1: Comparison: Placebo vs Tio R2.5; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.1114, Mixed Models Analysis; Adjusted using a restricted maximum likelihood (REML)-based mixed effects model with repeated measures (MMRM); Mean Difference (Final Values) = -0.953, 95% CI 2-sided [-2.125 to 0.220], Standard Error of Mean 0.598 — Tio R2.5 - Placebo
Statistical Analysis 2: Comparison: Placebo vs Tio R5; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.7665, Mixed Models Analysis; Adjusted using a restricted maximum likelihood (REML)-based mixed effects model with repeated measures (MMRM); Mean Difference (Final Values) = -0.178, 95% CI 2-sided [-1.355 to 0.999], Standard Error of Mean 0.600 — Tio R5 - Placebo

14. Secondary Outcome: Mean Pre-dose Morning FEV1 (FEV1 a.m.) Based on the Weekly Mean Response at Week 24
Description: as for outcome 11
Time Frame: Baseline and last 7 days before week 24 visit
Population: FAS
Measure: Mean (Standard Error); unit: Litre
Arm/Group | Placebo | Tio R2.5 | Tio R5 | Salmeterol
Number analyzed (Participants) | 235 | 238 | 236 | 247
Litre | 0.020 (0.023) | 0.099 (0.023) | 0.084 (0.023) | 0.103 (0.022)
Statistical Analysis 1: Comparison: Placebo vs Tio R2.5; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0111, Mixed Models Analysis; Adjusted using a restricted maximum likelihood (REML)-based mixed effects model with repeated measures (MMRM); Mean Difference (Final Values) = 0.079, 95% CI 2-sided [0.018 to 0.140], Standard Error of Mean 0.031 — Tio R2.5 - Placebo
Statistical Analysis 2: Comparison: Placebo vs Tio R5; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0395, Mixed Models Analysis; Adjusted using a restricted maximum likelihood (REML)-based mixed effects model with repeated measures (MMRM); Mean Difference (Final Values) = 0.064, 95% CI 2-sided [0.003 to 0.126], Standard Error of Mean 0.031 — Tio R5 - Placebo

15. Secondary Outcome: Mean Pre-dose Evening FEV1 (FEV1 p.m.) Based on the Weekly Mean Response at Week 24
Description: as for outcome 11
Time Frame: Baseline and last 7 days before week 24 visit
Population: FAS
Measure: Mean (Standard Error); unit: Litre
Arm/Group | Placebo | Tio R2.5 | Tio R5 | Salmeterol
Number analyzed (Participants) | 236 | 238 | 236 | 247
Litre | -0.002 (0.024) | 0.066 (0.023) | 0.064 (0.024) | 0.048 (0.023)
Statistical Analysis 1: Comparison: Placebo vs Tio R2.5; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0357, Mixed Models Analysis; Adjusted using a restricted maximum likelihood (REML)-based mixed effects model with repeated measures (MMRM); Mean Difference (Final Values) = 0.068, 95% CI 2-sided [0.005 to 0.131], Standard Error of Mean 0.032 — Tio R2.5 - Placebo
Statistical Analysis 2: Comparison: Placebo vs Tio R5; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0422, Mixed Models Analysis; Adjusted using a restricted maximum likelihood (REML)-based mixed effects model with repeated measures (MMRM); Mean Difference (Final Values) = 0.066, 95% CI 2-sided [0.002 to 0.129], Standard Error of Mean 0.032 — Tio R5 - Placebo

16. Secondary Outcome: Mean Number of Puffs of Rescue Medication During the Entire 24-h Day Based on the Weekly Mean Response at Week 24
Description: Daily use of salbutamol (albuterol) rescue medication as needed during the entire study period. Weekly means obtained during the last 7 days before week 24 measured by patients at home using the AM3 device. Response was defined as change from baseline. Means are adjusted for treatment, country, week, baseline, treatment by week, and baseline by week.
Time Frame: Baseline and last 7 days before week 24 visit
Population: FAS
Measure: Mean (Standard Error); unit: Number of Puffs
Arm/Group | Placebo | Tio R2.5 | Tio R5 | Salmeterol
Number analyzed (Participants) | 237 | 238 | 236 | 247
Number of Puffs | -0.952 (0.093) | -1.123 (0.092) | -0.843 (0.093) | -1.078 (0.091)
Statistical Analysis 1: Comparison: Placebo vs Tio R2.5; Analyses included the fixed, categorical effects of treatment, week, and treatment-by-week interaction, as well as the covariates of baseline value and baseline value-by-week interaction. Patient was included as a random effect in the model; Test type: Superiority or Other; p = 0.1927, Mixed Models Analysis; Adjusted using a restricted maximum likelihood (REML)-based mixed effects model with repeated measures (MMRM); Mean Difference (Final Values) = -0.171, 95% CI 2-sided [-0.427 to 0.086], Standard Error of Mean 0.131 — Tio R2.5 - Placebo
Statistical Analysis 2: Comparison: Placebo vs Tio R5; [analysis description as in outcome 16, analysis 1]; Test type: Superiority or Other; p = 0.4053, Mixed Models Analysis; Adjusted using a restricted maximum likelihood (REML)-based mixed effects model with repeated measures (MMRM); Mean Difference (Final Values) = 0.109, 95% CI 2-sided [-0.148 to 0.367], Standard Error of Mean 0.131 — Tio R5 - Placebo

17. Secondary Outcome: Asthma Symptom-free Days Based on the Weekly Mean Response at Week 24
Description: Weekly means obtained during the last 7 days before week 24 measured by patients at home using the AM3 device. Response was defined as change from baseline. Means are adjusted for treatment, country, week, baseline, treatment by week, and baseline by week. An asthma symptom-free day was defined as a day with no reported symptoms and no use of rescue medication.
Time Frame: Baseline and last 7 days before week 24 visit
Population: FAS
Measure: Mean (Standard Error); unit: Days
Arm/Group | Placebo | Tio R2.5 | Tio R5 | Salmeterol
Number analyzed (Participants) | 237 | 238 | 236 | 247
Days | 0.189 (0.023) | 0.164 (0.023) | 0.196 (0.023) | 0.195 (0.022)
Statistical Analysis 1: Comparison: Placebo vs Tio R2.5; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.3501, Mixed Models Analysis; Adjusted using a restricted maximum likelihood (REML)-based mixed effects model with repeated measures (MMRM); Mean Difference (Final Values) = -0.026, 95% CI 2-sided [-0.079 to 0.028], Standard Error of Mean 0.027 — Tio R2.5 - Placebo
Statistical Analysis 2: Comparison: Placebo vs Tio R5; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.8045, Mixed Models Analysis; Adjusted using a restricted maximum likelihood (REML)-based mixed effects model with repeated measures (MMRM); Mean Difference (Final Values) = 0.007, 95% CI 2-sided [-0.047 to 0.061], Standard Error of Mean 0.028 — Tio R5 - Placebo

18. Primary Outcome: The Responder Rate as Assessed by the ACQ From the Two Twin Trials 205.418 (NCT01172808) and the Present 205.419 (NCT01172821)
Description: The responder rate as assessed by the Asthma Control Questionnaire (ACQ) determined at the end of the 24-week treatment period (on combined data from the two twin trials 205.418 (NCT01172808) and 205.419 (NCT01172821)). A patient was considered to be a responder if he or she was reported with an improvement (decrease) in the ACQ total score of at least 0.5 points.
Time Frame: 24 weeks
Population: FAS of combined data from the two twin trials 205.418 (NCT01172808) and 205.419 (NCT01172821).
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Tio R2.5 | Tio R5 | Salmeterol
Number analyzed (Participants) | 518 | 515 | 513 | 535
Percentage of participants | 57.7 | 64.5 | 64.3 | 66.5
Statistical Analysis 1: Comparison: Placebo vs Tio R2.5; Test type: Superiority or Other; p = 0.0308, Fisher Exact — Calculated as 2*one-sided-p-value in the direction corresponding to testing the null hypothesis; Odds Ratio (OR) = 1.33, 95% CI 2-sided [1.03 to 1.72] — Tio R2.5 / Placebo
Statistical Analysis 2: Comparison: Placebo vs Tio R5; Test type: Superiority or Other; p = 0.0348, Fisher Exact — Calculated as 2*one-sided-p-value in the direction corresponding to testing the null hypothesis; Odds Ratio (OR) = 1.32, 95% CI 2-sided [1.02 to 1.71] — Tio R5 / Placebo

19. Secondary Outcome: Time to First Severe Asthma Exacerbation From the Two Twin Trials 205.418 (NCT01172808) and the Present 205.419 (NCT01172821)
Description: Time to first severe asthma exacerbation during the 24-week treatment period on combined data from the two twin trials 205.418 (NCT01172808) and 205.419 (NCT01172821)
Time Frame: 24 weeks
Population: FAS of combined data from the two twin trials 205.418 (NCT01172808) and 205.419 (NCT01172821)
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Placebo | Tio R2.5 | Tio R5 | Salmeterol
Number analyzed (Participants) | 518 | 515 | 513 | 535
weeks | NA [NA to NA] — The median time to first severe asthma exacerbation could not be calculated as less than 50% of patients in each treatment group experienced an asthma exacerbation. | NA [NA to NA] — The median time to first severe asthma exacerbation could not be calculated as less than 50% of patients in each treatment group experienced an asthma exacerbation. | NA [NA to NA] — The median time to first severe asthma exacerbation could not be calculated as less than 50% of patients in each treatment group experienced an asthma exacerbation. | NA [NA to NA] — The median time to first severe asthma exacerbation could not be calculated as less than 50% of patients in each treatment group experienced an asthma exacerbation.

20. Secondary Outcome: Time to First Asthma Exacerbation From the Two Twin Trials 205.418 (NCT01172808) and the Present 205.419 (NCT01172821)
Description: Time to first asthma exacerbation (including severe, non-severe; symptomatic, asymptomatic; i.e. any exacerbation) during the 24-week treatment period on combined data from the two twin trials 205.418 (NCT01172808) and 205.419 (NCT01172821)
Time Frame: 24 weeks
Population: FAS of combined data from the two twin trials 205.418 (NCT01172808) and 205.419 (NCT01172821)
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Placebo | Tio R2.5 | Tio R5 | Salmeterol
Number analyzed (Participants) | 518 | 515 | 513 | 535
weeks | NA [NA to NA] — The median time to first asthma exacerbation could not be calculated as less than 50% of patients in each treatment group experienced an asthma exacerbation. | NA [NA to NA] — The median time to first asthma exacerbation could not be calculated as less than 50% of patients in each treatment group experienced an asthma exacerbation. | NA [NA to NA] — The median time to first asthma exacerbation could not be calculated as less than 50% of patients in each treatment group experienced an asthma exacerbation. | NA [NA to NA] — The median time to first asthma exacerbation could not be calculated as less than 50% of patients in each treatment group experienced an asthma exacerbation.

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Placebo | Tio R2.5 | Tio R5 | Salmeterol
Serious Adverse Events (participants affected / at risk) | 4/254 | 7/257 | 7/253 | 4/266
Other Adverse Events (participants affected / at risk) | 102/254 | 89/257 | 87/253 | 90/266
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=254) | Tio R2.5 (N=257) | Tio R5 (N=253) | Salmeterol (N=266)
Anal fistula (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Ileus paralytic (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Suprapubic pain (General disorders) | 0 | 1 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0
Chemical poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Intestinal anastomosis complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 0
Cervicobrachial syndrome (Nervous system disorders) | 0 | 1 | 0 | 0
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Parovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1 | 1
Eosinophilic pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=254) | Tio R2.5 (N=257) | Tio R5 (N=253) | Salmeterol (N=266)
Nasopharyngitis (Infections and infestations) | 26 | 31 | 19 | 25
Upper respiratory tract infection (Infections and infestations) | 22 | 11 | 12 | 16
Peak expiratory flow rate decreased (Investigations) | 28 | 21 | 25 | 18
Asthma (Respiratory, thoracic and mediastinal disorders) | 54 | 44 | 50 | 52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.